CLINICAL TRIAL: NCT02314013
Title: Prospective Randomized Clinical Trial for the Management of Uncomplicated Diverticulitis in Right Colon; Non-antibiotics Versus Antibiotics
Brief Title: Randomized Clinical Trial for the Uncomplicated Diverticulitis in Right Colon
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dongtan Sacred Heart Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-023
Record Dates: First submitted 2014-11-20; First posted 2014-12-10 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-04

CONDITIONS: Simple Diverticular Disease
Keywords: uncomplicated diverticulitis, economic cost, hospital stay
MeSH Terms: interventions — Cephalosporins; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cephalosporin + Metronidazole (Active Comparator): intravenous antibiotics injection (3rd generation cephalosporin + metronidazole) and then change to oral antibiotics (3rd generation cephalosporin+ metronidazole) (an expected average 10 days)
  Interventions: Drug: Cephalosporin + Metronidazole
- No antibiotic (No Intervention): bowel rest and then, discharge until tolerable soft diet.

INTERVENTIONS:
Drug: Cephalosporin + Metronidazole — intravenous antibiotics injection (3rd generation cephalosporin + metronidazole)and then change to oral antibiotics (3rd generation cephalosporin+ metronidazole) (an expected average 10 days)
  Arms: Cephalosporin + Metronidazole

SUMMARY:
The aim of the present study was to evaluate whether antibiotics is mandatory for the treatment of acute uncomplicated right-sided diverticulitis.

The hypothesis is that patients having acute uncomplicated diverticulitis at right-sided colon will be recovered without antibiotics.

DETAILED DESCRIPTION:
All patients in the study were randomly allocated to one of the following two treatment groups; no-antibiotics group or antibiotics group.

Patients of no-antibiotics group were admitted to the ward and administered intravenous fluid and bowel rest at least up to 5 days until clinical symptom and sign were stabilized. And then the patient discharge until oral intake was tolerated.

In antibiotics group, the treatment was initiated with an intravenous combination of a third generation cephalosporin or quinolone and metronidazole until oral intake was tolerated. Oral antibiotics such as cefpodoxime together with metronidazole were initiated subsequently on the ward. The total duration of antibiotic treatment was an expected average 10days.

Patients in both group were re-visited outpatient clinic after an expected average 7 days for check-up of serology test (including complete blood count and C-reactive protein), and after an expected average 6 weeks for CT. If the patients did not re-visit outpatient clinic, we checked the call.

ELIGIBILITY:
Inclusion Criteria:

* Right-sided colonic diverticulitis
* Uncomplicated diverticulitis

Exclusion Criteria:

* Pregnancy
* Refuse to investigation
* Immunosuppressive therapy or immunologic incompetence
* Colonic diverticulitis except right-sided diverticulitis
* Complicated diverticulitis
* Disorder of psychology or cognition
* Allergic reaction to antibiotics being used in the study (3rd generation cephalosporin, quinolone, metronidazole)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-11 (Actual); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Treatment Failure | 4-6 weeks
  advancement or recurrence diverticulitis at the same site.

SECONDARY OUTCOMES:
length of hospital stay at first admission for diverticulitis | up to 2 weeks
total cost of hospitalization for diverticulitis | up to 2 weeks
  length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Jong Wan Kim, MD, Principal Investigator — Department of Surgery, Dongtan Sacred Heart Hospital, Hallym University College of Medicine
Locations (1):
- Department of Surgery, Dongtan Sacred Heart Hospital, Hallym University College of Medicine, Hwaseong-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kim JY, Park SG, Kang HJ, Lim YA, Pak KH, Yoo T, Cho WT, Shin DW, Kim JW. Prospective randomized clinical trial of uncomplicated right-sided colonic diverticulitis: antibiotics versus no antibiotics. Int J Colorectal Dis. 2019 Aug;34(8):1413-1420. doi: 10.1007/s00384-019-03343-w. Epub 2019 Jul 2. PMID 31267222